CLINICAL TRIAL: NCT00339118
Title: EpSSG (European Soft Tissue Sarcoma Study Group) Protocol for Non-Metastatic Rhabdomyosarcoma in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SHEBA-06-4013-IK-CTIL
Record Dates: First submitted 2006-06-19; First posted 2006-06-20 (Estimated); Last update posted 2006-06-20 (Estimated); Status verified 2006-06

CONDITIONS: Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: doxorubicin, cytoxan

SUMMARY:
The purpose of the study is achieve standardization treatment of low and intermediate risk rhabdomyosarcoma patients, with an attempt to improve treatment results in high and very high risk patients by the addition of doxorubicin as induction treatment and at the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* child
* non metastatic rhabdomyosarcoma
* adequate heart, kidney, liver function

Exclusion Criteria:

* age over 21 years, under 6 months
* metastatic disease
* heart, kidney, liver disease

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

PRIMARY OUTCOMES:
event free survival
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Iris Kventsel, MD, Principal Investigator — Sheba Medical Center

REFERENCES:
- [Derived] Bisogno G, Chisholm J, Hladun R, De Salvo GL, Guerin F, Casanova M, Mandeville H, Alaggio R, Coppadoro B, Orbach D, Ferrari A, van Rijn R, Defachelles AS, Ben-Arush M, Glosli H, Cesen M, Merks JHM, Minard-Colin V. Maintenance Chemotherapy in Patients With High-Risk Rhabdomyosarcoma: Long-Term Survival Analysis of the European Paediatric Soft Tissue Sarcoma Study Group RMS 2005 Trial. J Clin Oncol. 2025 Jun;43(16):1856-1862. doi: 10.1200/JCO-24-02850. Epub 2025 Mar 7. PMID 40053891
- [Derived] Bisogno G, Minard-Colin V, Zanetti I, Ferrari A, Gallego S, Davila Fajardo R, Mandeville H, Kelsey A, Alaggio R, Orbach D, Terwisscha van Scheltinga S, Guillen Burrieza G, Ben-Arush M, Glosli H, Mudry P, Ferman S, Devalck C, Defachelles AS, Merks JHM, Jenney M. Nonmetastatic Rhabdomyosarcoma in Children and Adolescents: Overall Results of the European Pediatric Soft Tissue Sarcoma Study Group RMS2005 Study. J Clin Oncol. 2023 May 1;41(13):2342-2349. doi: 10.1200/JCO.22.02093. Epub 2023 Feb 27. PMID 36848614
- [Derived] Bisogno G, De Salvo GL, Bergeron C, Gallego Melcon S, Merks JH, Kelsey A, Martelli H, Minard-Colin V, Orbach D, Glosli H, Chisholm J, Casanova M, Zanetti I, Devalck C, Ben-Arush M, Mudry P, Ferman S, Jenney M, Ferrari A; European paediatric Soft tissue sarcoma Study Group. Vinorelbine and continuous low-dose cyclophosphamide as maintenance chemotherapy in patients with high-risk rhabdomyosarcoma (RMS 2005): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2019 Nov;20(11):1566-1575. doi: 10.1016/S1470-2045(19)30617-5. Epub 2019 Sep 24. PMID 31562043